CLINICAL TRIAL: NCT02743559
Title: Does Antenatal Vitamin D Supplementation Influence Bone's Postnatal Response to Mechanical Stimulation?
Brief Title: Does Vitamin D Alter Bone's Response to Vibration?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); University of Southampton (Other); University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCH/15/094
Record Dates: First submitted 2016-04-05; First posted 2016-04-19 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Vitamin D Deficiency; Osteoporosis
MeSH Terms: conditions — Vitamin D Deficiency; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D group (Active Comparator): Children born to mothers who received vitamin D during pregnancy will undergo mechanical stimulation using whole body vibration(WBV) by standing on the vibration platform(LivMd) for 10 minutes on 5 consecutive mornings, at 7.30-8 am.
  Interventions: Device: Mechanical Stimulation using whole body vibration
- Placebo group (Placebo Comparator): Children born to mothers who received placebo during pregnancy will also undergo mechanical stimulation using whole body vibration(WBV) by standing on the vibration platform (LivMd) for 10 minutes on 5 consecutive mornings, at 7.30-8 am.
  Interventions: Device: Mechanical Stimulation using whole body vibration

INTERVENTIONS:
Device: Mechanical Stimulation using whole body vibration — All participants will undergo whole body vibration (WBV) by standing on the LivMD WBV platform on 5 consecutive mornings

SUMMARY:
Fractures in children are common and the incidence is increasing. They are more common in children who have small, narrow and weak bones. Studies have shown that fractures in early childhood are associated with later bone strength.

There are several (i) non-modifiable (age, gender, race, genetics) and (ii) modifiable factors such as nutrition (vitamin D & calcium intake) and exercise that can contribute to bone strength.

Low calcium is associated with an increased risk of fracture. Vitamin D plays a pivotal role in bone health by increasing the absorption of calcium from the gut. Investigators know from the previous research that there is a reduction in bone strength in children whose mothers had lower vitamin D levels during pregnancy.

Bone growth can also be achieved by loading of bone during childhood in the form of regular sport activities such as gymnastics and exercise programmes. Equally it can be achieved by using whole body vibration (WBV). WBV is the application of vibratory stimulus to the body in a synchronous fashion by which the bones are made much stronger reducing the risk of fracture in later life. Thus WBV can be used as a means to assess bone responsiveness to mechanical stimulation. Studies have shown that standing on a vibrating platform for 10 minutes a day can significantly increase the bone mass. Investigators' own research has also shown that healthy boys when made to stand on a vibration platform for 10 minutes daily for 5 days increased the strength and quality of their bones.

Thus the role of diet and mechanical loading are of considerable interest in determining their role in bone health and the prevention of fractures.

Maternal Vitamin D Osteoporosis Study (MAVIDOS) is a large study conducted recently at 3 different big centres (Sheffield, Southampton and Oxford). Results from this study have shown that giving a higher dose of vitamin D to pregnant women every day from 14 weeks of pregnancy increased the strength of the bones in their infants. In the proposed study Investigators aim to show how vitamin D supplementation during pregnancy affects the response of bone to vibration in children whose mothers participated in the MAVIDOS study in Sheffield. These children will be 4 years of age when they participate in this study.

The results of this study will help inform public health policy on vitamin D intake during pregnancy. This will also help the investigators identify a possible risk factor for poor bone health in children.

DETAILED DESCRIPTION:
This project aims to determine whether antenatal vitamin D supplementation alters postnatal bone formation in response to mechanical stimulation.

The skeleton responds to mechanical stimulation by an increase in bone size and mass and that increment can persist into adult life and may lower the risk of osteoporosis (Daly, & Bass, 2009). In contrast, without mechanical stimulation, bone is lost.

Cells within bone - osteoblasts and osteoclasts - are involved in the removal and formation of bone; the biomarkers Pro-collagen type 1 N-terminal propeptide (PINP) and C-terminal cross-linked telopeptide of type I collagen (CTx) are surrogates for their respective tissue level activities.

Whole body vibration (WBV) has been used as one of the methods to deliver mechanical stimulation in both adults and children.

The investigators have recently shown in healthy boys aged 9-11 years, WBV experienced 10 minutes daily for five days increases the P1NP by 25% and CTx by 11% (Harrison et al., 2015).

The investigators undertook another study recently to determine the effect of reduced vitamin D intake during pregnancy and early life on the skeleton's response to mechanical loading using a mouse model.

Our unpublished data show that antenatal vitamin D depletion substantially reduces the loading-dependent increase in both cortical and trabecular bone mass of offspring mice close to skeletal maturity.

The available human and mouse data suggest that antenatal vitamin D deficiency in some way influences the bone to become less responsive to mechanical stimulation.

The investigators are now ready to explore this in humans, to assess the responsiveness of the skeleton to mechanical stimulation by using WBV in the children who have been exposed to higher levels of vitamin D in-utero through maternal supplementation of vitamin D.

Through this study the investigators will be able to determine whether the in-utero environment can be modified easily to improve the skeletal responsiveness to activity and this improved skeletal health in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* All children born to mothers who participated in MAVIDOS trial in Sheffield free from any condition affecting bone health, general nutrition, growth and glucose metabolism will be invited to enrol in the study.

Exclusion Criteria:

* Children with (1) balance problems, (2) current or healing fractures (3) any chronic illness involving the bone, liver and kidney (4) current long-term use of steroids, anticonvulsants or any medication that might affect calcium and vitamin D metabolism will be identified from through a questionnaire and excluded.
* Participants will fill in questionnaires to estimate their calcium intake and Vitamin D exposure and this will be included in the analysis

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Difference in mean increase in the bone turnover marker Pro-collagen type 1 N-terminal propeptide (P1NP) between children born to antenatally vitamin D replete mothers versus antenatally vitamin D deficient mothers. | 2 years

SECONDARY OUTCOMES:
Change in C-terminal cross-linked telopeptide of type I collagen(CTx) | 2 years
Change in Osteoprotegerin(OPG). | 2 years
Change in parathyroid hormone (PTH). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sujatha Gopal, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided